CLINICAL TRIAL: NCT00433043
Title: Beta-blocker Uptitration in Heart Failure Patients Receiving Cardiac Resynchronization Therapy With Optivol Fluid Status Monitoring System
Brief Title: BOAT: Beta Blocker Uptitration With OptiVol After Cardiac Resynchronization Therapy (CRT)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-107
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2014-01

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; Beta blockers; Resynchronization; Congestive Heart Failure, NYHA III-IV; Candidate for BIVPM; Not on Target Dose (Coreg 25 Bid or Toprol XL 200 qd)
MeSH Terms: conditions — Heart Failure | interventions — Adrenergic beta-Antagonists; Carvedilol; Metoprolol; Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CRT and b-blocker uptitration to target dose
  Interventions: Drug: Beta blocker (carvedilol or metoprolol succinate); Procedure: CRT (cardiac resynchronization therapy)
- 2 (Active Comparator): CRT and continuation of entry b-blocker dose to 6 month evaluation
  Interventions: Drug: Beta blocker (carvedilol or metoprolol succinate); Procedure: CRT (cardiac resynchronization therapy)

INTERVENTIONS:
Drug: Beta blocker (carvedilol or metoprolol succinate) — Both groups get CRT. Group 1 is uptitrated to target dose beta blocker after CRT. Group 2 maintains their b-blocker dose from study entry.
Procedure: CRT (cardiac resynchronization therapy) — Both arms

SUMMARY:
Many heart failure patients are unable to reach target beta blocker doses. This study will address whether cardiac resynchronization therapy (CRT) will enable uptitration of beta-blockers to target doses and whether it will favorably affect remodeling by reducing left ventricular end systolic volume (LVESV), with measurable clinical benefit, beyond CRT alone (without changes in beta-blocker dose).

DETAILED DESCRIPTION:
Beta blockers have been proven to have benefit in heart failure (HF) patients with regard to morbidity and mortality. However, initiation and uptitration remains a challenge in many patients. Worsening of heart failure, symptomatic hypotension and symptomatic bradycardia all limit up-titration to the target doses that have been shown to have mortality benefits (carvedilol [Coreg] 25 mg bid, metoprolol succinate [Toprol-XL] 200 mg qd) in the large clinical trials (COPERNICUS, MERIT-HF).

It is debated whether the benefit of beta-blockade is solely due to heart rate reduction or more broadly from the cardiac, central and peripheral effects of blocking sympathetic activity. Clearly, there is a remodeling effect on the dilated ventricle. Furthermore, patients with heart rates of 64 bpm or less are rarely begun on beta-blocker therapy. It is not known whether these patients should be given a pacemaker in order to then safely initiate beta-blocker therapy.

It is also clear that isolated right ventricular pacing can have deleterious effects on ventricular dyssynchrony and symptomatic heart failure despite medical therapy. Biventricular pacing (BIVPM), also known as cardiac resynchronization therapy (CRT), is the pacing mode of choice for patients with wide QRS complexes and symptomatic HF.

It is hypothesized that CRT therapy allows for increased Beta -blocker dose (or initiation of beta-blocker in patients previously intolerant) with improved NYHA, ejection fraction, and remodeling effects. The synergy between two established heart failure therapies requires further evaluation in a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* NYHA III-IV
* QRS > 120 msec
* On medical therapy, but beta blocker dose not @ target (carvedilol 25 bid, metoprolol succinate 200 qd)

Exclusion Criteria:

* QRS < 120 msec
* On target beta blocker dose

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
LVESVI change in patients with CRT/ increased dose of beta-blockers vs CRT and no change in beta-blocker dose. | 6 months

SECONDARY OUTCOMES:
Correlation of Optivol fluid measurement increases (decreased impedance) with symptomatic worsening of heart failure during beta blocker uptitration | 6 months
Optivol measurements (decreased impedance, increase volume index) correlated with the need for adjusting diuretic therapy when uptitrating beta blocker dose | 12 months
Functional improvements | 6 months
Exercise - 6 minute walk | 6 months
QOL - NYHA, Minnesota LWHFQ, Symptom Assessment Questionnaire | 6 months
Ejection fraction | 6 months
LVEDVI | 6 months
Remodeling | 6 months
HF Hospitalizations/ Mortality | 6 months
Evaluation of LVESVI in patients who actually achieve target dose | 6 months
Comparison of LVESVI changes based on initial beta-blocker dose | 6 months
Plasma Brain natriuretic peptide (BNP) change | 6 months
12 month comparison after Group 2 has been uptitrated. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marrick L Kukin, MD, Principal Investigator — St. Luke's Roosevelt Hospitals
Locations (3):
- United States (3):
  - St. Lukes Roosevelt Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Jefferson Medical College, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Aranda JM Jr, Woo GW, Conti JB, Schofield RS, Conti CR, Hill JA. Use of cardiac resynchronization therapy to optimize beta-blocker therapy in patients with heart failure and prolonged QRS duration. Am J Cardiol. 2005 Apr 1;95(7):889-91. doi: 10.1016/j.amjcard.2004.12.023. PMID 15781026
- [Background] Effect of metoprolol CR/XL in chronic heart failure: Metoprolol CR/XL Randomised Intervention Trial in Congestive Heart Failure (MERIT-HF). Lancet. 1999 Jun 12;353(9169):2001-7. PMID 10376614
- [Background] Packer M, Coats AJ, Fowler MB, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Castaigne A, Roecker EB, Schultz MK, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival Study Group. Effect of carvedilol on survival in severe chronic heart failure. N Engl J Med. 2001 May 31;344(22):1651-8. doi: 10.1056/NEJM200105313442201. PMID 11386263
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059